CLINICAL TRIAL: NCT07052838
Title: A Multicenter, Single-Arm, Open-Label Phase III Clinical Study Evaluating the Efficacy and Safety of HSK39297 Tablets in Paroxysmal Nocturnal Hemoglobinuria Patients With Anemia Despite Stable Anti-C5 Antibody Therapy
Brief Title: Efficacy and Safety of HSK39297 in Anti-C5 Treated PNH Patients With Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK39297-302
Record Dates: First submitted 2025-06-29; First posted 2025-07-07 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Nocturnal Haemoglobinuria (PNH)
Keywords: Paroxysmal Nocturnal Hemoglobinuria
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSK39297 (Experimental)
  Interventions: Drug: HSK39297 tablets

INTERVENTIONS:
Drug: HSK39297 tablets — 200mg QD

SUMMARY:
The purpose of this study is to evaluate the efficacy of HSK39297 tablets in paroxysmal nocturnal hemoglobinuria (PNH) patients with anemia after stable treatment of anti-C5 antibody.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years, Male and female patients.
* Diagnosis of PNH based on flow cytometry showing >10% granulocyte clone size during the screening period.
* Stable use of Anti-C5 antibody at least 6 months prior to enrollment.
* Hemoglobin level < 10 g/dL at screening.

Exclusion Criteria:

* Hereditary or acquired complement deficiency.
* Active primary or secondary immunodeficiency.
* History of splenectomy, bone marrow/hematopoietic stem cell or solid organ transplants.
* History of recurrent invasive infections caused by encapsulated organisms( e.g. meningococcus or pneumococcus) or Mycobacterium tuberculosis.
* Patients with laboratory evidence of bone marrow failure (reticulocytes < 100x109/L, or platelets < 30x109/L or neutrophils < 0.5x109/L).
* Active systemic infection within 2 weeks prior to study drug administration.
* History of serious comorbidities that have been determined to be unsuitable for participation in the study.
* Pregnant or Lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2026-01-05 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving hemoglobin levels ≥ 120 g/L at least on three out of four measurements in the absence of red blood cell transfusions | 18 to 24 weeks

SECONDARY OUTCOMES:
Proportion of participants with increase in hemoglobin levels from baseline of ≥20 g/L at least on three out of four measurements in the absence of red blood cell transfusions | 18 to 24 weeks
Percentage of patients who did not receive a blood transfusion. | 18 to 24 weeks
Change from baseline in hemoglobin | Baseline, week 18 to 24
Change From Baseline in Reticulocyte Count | Baseline, week 18 to 24
Change from baseline in Functional Assessment of Chronic Illness Therapy (FACIT) - Fatigue score | Baseline, week 18 to 24
  The FACIT-F is a 13-item questionnaire with a 0-52 range. A higher total score indicates less fatigue and better function.
Percent change from baseline in lactate dehydrogenase (LDH) | Baseline, week 18 to 24
Rate of breakthrough hemolysis (BTH) | 24 weeks
Proportion of participants with Major Adverse Vascular Events (MAVEs) | 24 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No